CLINICAL TRIAL: NCT05013372
Title: A Pioneering Study on the Safety and Efficacy of CD147-Chimeric Antigen Receptor (CAR) T Cells in Patients With Relapsed or Refractory T-cell Non-Hodgkin's Lymphoma
Brief Title: CD147-CAR T Cells for Relapsed/Refractory T Cell Non-Hodgkin's Lymphoma
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao-Jun Huang, Prof., Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD147-CAR T for R/R T-NHL
Record Dates: First submitted 2021-08-16; First posted 2021-08-19 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-08

CONDITIONS: T-cell Non-Hodgkin's Lymphoma
Keywords: CAR T cells; T-cell Non-Hodgkin's lymphoma; CD147
MeSH Terms: conditions — Lymphoma, T-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose-escalation (Other): Dose -1：0.1×10E+6/kg Dose 1：0.25×10E+6/kg Dose 2：0.5×10E+6/kg Dose 3：1.0×10E+6/kg Dose 4：2.0×10E+6/kg
  Interventions: Drug: CD147- CAR T cells

INTERVENTIONS:
Drug: CD147- CAR T cells — CAR T cells targeting CD147
  Other Names: CAR T cells targeting CD147

SUMMARY:
The safety and preliminary effectiveness of CD147-CAR T cells in patients with relapsed or refractory T cell non-Hodgkin's lymphoma will be investigated in this pioneering study.

DETAILED DESCRIPTION:
CD147 has been demonstrated higher and relatively specific expression on T cell non-Hodgkin's lymphoma. Preclinical studies have shown that CAR T cells targeting CD147 antigen can continuously eliminate Jurkat T-cell lymphoma in mice and extend survival without severe adverse events including hemolysis. Preliminary investigation of CD147-CAR T cells in solid tumors has started and shown an acceptable safety profile. The safety and preliminary effectiveness of CD147-CAR T cells in patients with relapsed or refractory T cell non-Hodgkin's lymphoma will be investigated in this pioneering study.

ELIGIBILITY:
Inclusion Criteria:

* The subject must meet all of the following criteria:

  1. 18-65 years old;
  2. Relapsed or refractory T-NHLs, including peripheral T-cell lymphoma, not otherwise specified (PTCL-NOS), angioimmunoblastic T-cell lymphoma (AITL), ALK-positive ALCL, ALK-negative Image result for anaplastic large cell lymphoma (ALCL), enteropathy-related T-cell lymphoma, hepatosplenic T-cell lymphoma, etc.;
  3. Previously received ≥2 lines of treatment without a complete response;
  4. Immunohistochemical detection of tumor cells CD147 positive;
  5. ECOG score 0-2;
  6. The collection of mononuclear cells can be performed upon the judgment of the researcher;
  7. No contraindications for allogeneic hematopoietic stem cell transplantation (AlloHCT);
  8. Have donors for AlloHCT;
  9. Agree for sequential treatment of AlloHCT;
  10. Without serious organ dysfunction in 2 weeks before CAR-T infusion:

      1. Heart: without arrhythmia, LVEF≥50%, and without pericardial effusion; without heart failure (NYHA class III or IV) within12 months before CAR-T infusion; without myocardial infarction within 12 months before CAR-T infusion; without long-QT syndrome or secondary QT interval prolongation;
      2. Liver: ALT<2 times the upper limit of normal (ULN) and TBIL<1.5 times ULN, without active hepatitis;
      3. APTT and PT<1.5 times ULN;
      4. Kidney: Serum creatinine <1.5 mg/dl; or if the serum creatinine exceeds the upper limit, eGFR (CKD-EPI formula) needs to be > 50 ml/min;
      5. Fingertip blood oxygen saturation ≥ 92%.
  11. Estimated survival ≥ 3 months;
  12. Sexually active patients must be willing to use an effective method of birth control during the study period and within 6 months after the study ending, and male partners should use condoms;
  13. The patient is willing to join this clinical trial and sign an informed consent.

Exclusion Criteria:

* Anyone who has one or more of the following:

  1. A history of other malignancies with a disease-free period < 5 years (except for cured basal cell carcinoma of the skin, cured cervical carcinoma in situ, and gastrointestinal tumors proven to be cured by endoscopic mucosal resection);
  2. Those who have received allogeneic hematopoietic stem cell transplantation or organ transplantation;
  3. Patients with bone marrow involvement;
  4. Those who are allergic to the biological agents in CAR-T cell product ;
  5. Pregnant or breastfeeding;
  6. Active bacterial, fungal or viral infection;
  7. Receiving systemic hormone therapy 1 week before participating in the clinical trial;
  8. Have received other gene therapy before;
  9. HBV or HCV infection or carrier is defined as: HBsAg positive or HBV-DNA positive; anti-HCV positive and HCV-RNA positive;
  10. Active HIV infection;
  11. Clinical diagnosis of virus infection or uncontrolled virus activation, including cytomegalovirus (CMV), adenovirus (ADV), BK virus or human herpesvirus 6 (HHV-6), etc.;
  12. Central nervous system lymphoma (CNSL) is defined as the presence of ≥5 tumor cells/ ul in cerebrospinal fluid (CSF) or MRI suggested CNSL; any other CNS diseases, such as uncontrolled epilepsy, cerebral ischemia/hemorrhage, dementia, cerebellar disease or any autoimmune disease involving the central nervous system, or received treatment for central nervous system or brain metastasis (radiotherapy, surgery or other treatments);
  13. Imaging determined lung infection;
  14. Inappropriate to participate in the trial with investigators' decision.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | within 12 months
  The highest dose that does not cause unacceptable side effects.
Dose-limiting toxicity (DLT) | within 12 months
  Side effects serious enough to prevent an increase in dose.
Adverse events | within 12 months
  Adverse events
Serious adverse events (SAE) | within 12 months
  Serious adverse events (SAE)
Adverse events of special interest (AESI) | within 12 months

SECONDARY OUTCOMES:
Overall response rate (ORR) | At the 12th week, 6th month, 9th month and 12th month
  Overall response rate (ORR) evaluated according to the Lugano2014 criteria
Complete response rate (CR) | At the 12th week, 6th month, 9th month and 12th month
  Complete response rate (CR) evaluated according to the Lugano2014 criteria
Duration of response (DOR) | At the 12th week, 6th month, 9th month and 12th month
  Duration of response (DOR)
Cmax of CD147-CAR T cells | within 4 weeks
Tmax of CD147-CAR T cells | within 4 weeks
AUC of CD147-CAR T cells | within 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojun Huang, MD. PhD., Principal Investigator — Peking University People's Hospital

IPD SHARING:
Plan to Share IPD: No